CLINICAL TRIAL: NCT04655560
Title: Understanding Barriers and Facilitators to the Participation of Women Living With HIV in Clinical Trials : a Mixed-method Study (EVA)
Acronym: EVA
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Principal Investigator, Calmy Alexandra, Professor, University Hospital, Geneva
Other Study IDs: 2020-02286
Record Dates: First submitted 2020-11-13; First posted 2020-12-07 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: HIV
Keywords: HIV; Clinical trials; Women; qualitative study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women living with HIV
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — qualitative study

SUMMARY:
To identify the most important barriers and facilitators to the participation of cisgender women living with HIV in clinical trials (perceived and real) and to establish possible mechanisms leading to refusal of trial participation. Specifically, psychosocial factors and/or cultural environments that enhance or undermine HIV-positive cisgender women's participation. These can include social inclusion, confidence in research, perceived personal vulnerability, cultural, familial and professional environment.

The investigators expect to propose pragmatic solutions to enhance participation of HIV-positive cisgender women in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women
* Adult (>18 years) HIV-infected
* Informed consent documented by signature
* Patients under stable antiretroviral therapy
* French speaking (sufficient fluency for a conversation)

Exclusion Criteria:

* Having participated in a previous qualitative study about Cure Trials acceptability among HIV patients
* Incapable of discernment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women living with HIV
  Note: ethnicity will not represent a selection's criteria. However, special care will be payed to assure a certain heterogeneity in the sample concerning this aspect.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of barriers and facilitators to the participation of women in clinical trials (HIV) through a questionnaire | through study completion, an average of 1 year
  Specific questions will be asked during a face-to-face interview to identify factors favoring or barriers to the participation of women in clinical trials.
Evaluation of mechanisms leading to refusal of trial participation through a questionnaire | through study completion, an average of 1 year
  Specific questions will be asked during a face-to-face interview to understand mechanisms leading to refusal of trial participation.
  Specifically, psychosocial factors and/or cultural environments that enhance or undermine HIV-positive cisgender women's participation. These can include social inclusion, confidence in research, perceived personal vulnerability, cultural, familial and professional environment.

SECONDARY OUTCOMES:
Offering solutions for a better inclusion of HIV-women in clinical trials - qualitative study | through study completion, an average of 1 year
  Analysis of questionnaires allowing recommendations to be made

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No